CLINICAL TRIAL: NCT00812032
Title: Evaluation of Antiplatelet Effects of Different Dosages of Aspirin in Type 2 Diabetic Patients
Acronym: DM-ASA 001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Paul Hjemdahl, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EudraCT No: 2007-003186-40
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: NIDDM; Aspirin; platelet inhibition; Aspirin treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aspirin — 75 mg per day versus 75 mg twice daily and 320mg once daily
  Other Names: Trombyl
Drug: aspirin — crossover study with three dosages: 75 mg once daily, 75 mg twice daily, 320 mg once daily.
  Other Names: Trombyl

SUMMARY:
The efficacy of low dose aspirin appears to be substantially lower in diabetic patients, compared to patients without diabetes. The aim of the investigators study is to test the laboratory response to different dosing of aspirin in type 2 Diabetes Mellitus. The investigators will compare the regular dose of 75mg once daily to 75 mg twice daily or to 320 mg once daily. The hypothesis of the study is that twice daily dosing of aspirin may improve the response to aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM with micro- or macroangiopathy.
* HbA1c 6-9 % (Mono-S method).
* Need for, or already on-going aspirin treatment.
* Age 50-75 years
* Antecubital forearm veins allowing technically good sampling for platelet studies

Exclusion Criteria:

* Diet controlled DM.
* Acute ischemic stroke, acute coronary syndrome, (myocardial infarction or unstable angina pectoris), or revascularization by PCI or by-pass surgery within the last 6 months.
* Acute or chronic kidney disease (P-cystatin C within the reference interval)
* Acute or chronic liver disease (ALAT ≤2 times the upper reference value).
* A history of gastric or duodenal ulcer disease.
* Need for treatment with anticoagulants, clopidogrel, NSAID's, or thiazolidinediones.
* Thrombocytopenia (platelet count <150 x 109/L)
* Anticipated need for alteration of concomitant drug therapy during the course of the study.
* Enrollment in another clinical study.
* Contraindication(s) to aspirin treatment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
An exploratory study with three co-primary response variables which are directly related to platelet COX-1 inhibition: arachidonic acid-induced platelet aggregation in whole blood and PRP and in the Cone-and-Plate(let) Assay (CPA) | 12 or 24 hours after last dose of Aspirin

SECONDARY OUTCOMES:
Indirectly COX-related platelet aggregation induced by collagen or ADP, and thromboxane metabolite excretion. | 12 or 24 hours after last dose of aspirin

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hjemdahl, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Medicine, Clinical pharmacology Unit, Karolinska University Hospital, Solna., Stockholm, Sweden